CLINICAL TRIAL: NCT03001518
Title: Immunologic Signatures Following Surgery for Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00077435
Record Dates: First submitted 2016-12-15; First posted 2016-12-23 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer; Surgery
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma from 4 blood draws
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery: No intervention. Patients who undergo surgical resection of their pancreatic cancer.

SUMMARY:
The goal of this pilot study is to evaluate and describe the immunologic and overall outcomes of subjects who undergo routine pancreatectomy with or without irreversible electroporation (IRE) for pancreatic cancer. Immunologic markers in the blood will be measured at several time points before and after surgery to determine if surgical approach is associated with different immunologic responses. Secondary outcomes will include mortality and morbidity; operative time; blood loss and transfusion requirements; and oncologic outcomes such as: margin status, lymph node harvest, disease-free survival, and overall survival. Analysis of immune response will help the investigator determine whether to expand the pilot into a larger study.

DETAILED DESCRIPTION:
Subjects will have blood draws at the following timepoints: Pre-op, 1-2 days post-op, 3-5 days post-op, and 1-4 months post-op. At each timepoint, three 8.5mL ACD (yellow top) vacutainer tubes will be drawn by the Biobank and Translational Research Core (BRTC), study personnel, or hospital phlebotomists. The blood will be processed for PBMC isolation by BRTC for Dr. Weinhold's laboratory and will be viable within 8 hours of draw. These timepoints for blood draws are at the same time as usual operative care and will not require additional visits on the part of the subject.

For this study we will extensively utilize several polychromatic flow cytometry (PFC) platforms to follow activation, maturation, exhaustion, and proliferation patterns within CD4+ and CD8+ subsets of T-cells. We will also utilize an intracellular cytokine staining (ICS) platform in efforts to detect anti-tumor associated antigen (TAA) responses by CD4+ and CD8+ T cells from peripheral blood mononuclear cells (PBMC) as well as lymphocytes infiltrating the patient's tumor. These assays are designed to measure antigen-driven intracellular production of IFN-γ, TNF-α, and IL-2, as well as the degranulation marker CD107. This strategy enables us to not only document individual cytokine responses, but to also assess (through Boolean gating) changes in relative polyfunctionality of the responses.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age and at least the minimum age of majority according to applicable State or Country Law.
* Subject is a suitable surgical candidate, i.e., is able to undergo general anesthesia and pancreatectomy for diagnosis of cancer
* Subject is willing and able to undergo additional blood draws

Exclusion Criteria:

• Subject is not a suitable candidate for surgery, or surgery is unable to be completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic ductal adenocarcinoma who undergo surgical resection of the cancer, with or without irreversible electroporation.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
immune response | preoperatively to 3 months postoperatively
  proliferation of immune cells in peripheral plasma

SECONDARY OUTCOMES:
90-day mortality | 90 days
  death by 90 days
surgical-site infection (SSI) | 90 days
  occurrence of superficial or deep infection of incision(s), by erythema/warmth/pain/swelling, need for antibiotics, positive wound cultures, purulent drainage/abscess, need to open skin incision, fascial dehiscence, etc. or documentation in the record of SSI. Organ/space infection indicated by abscess, anastomotic dehiscence, positive culture, etc. or documentation in the record of same.
pancreatic leak by qualitative appearance or amylase level | 90 days
  Drain output or CT-guided drainage consistent with pancreatic fluid in appearance and/or amylase level, or documentation in record of same.
operative time | 1 day
  time from start to end of operation
use of neoadjuvant therapy | 1 day
  used = 1
use of adjuvant therapy | 90 days
  used = 1
CA 19-9 level | 90 days
  result
return to operating room | 90 days
  Reoperation for exploration or repair of complication of primary procedure. Does not include wound debridement, placement of inferior vena cava filter, interventional radiology procedures, or other procedures unrelated to the initial procedure.
Non-SSI infection | 90 days
  Any infection not covered by surgical-site infection, such as urinary tract infection or pneumonia.
margin status | 1 week
  clean or unclean
intraoperative transfusion | 1 day
  used = 1
lymph node status | 1 week
  positive or negative
overall survival | 5 years
  number of months alive
disease-free survival | 5 years
  number of months without disease

CONTACTS AND LOCATIONS:
Overall Officials: Sabino Zani, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No